CLINICAL TRIAL: NCT00655655
Title: A Phase I Trial of the mTOR Inhibitor RAD001 in Combination With VEGF Receptor Tyrosine Kinase Inhibitor PTK787/ZK 222584 in Patients With Advanced Solid Tumors
Brief Title: Everolimus and Vatalanib in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0414; NCI-2009-01200 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC0414 (Other: Mayo Clinic)
Record Dates: First submitted 2008-04-09; First posted 2008-04-10 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Gastrinoma; Glucagonoma; Insulinoma; Metastatic Gastrointestinal Carcinoid Tumor; Metastatic Pheochromocytoma; Pancreatic Polypeptide Tumor; Recurrent Gastrointestinal Carcinoid Tumor; Recurrent Islet Cell Carcinoma; Recurrent Melanoma; Recurrent Neuroendocrine Carcinoma of the Skin; Recurrent Non-small Cell Lung Cancer; Recurrent Pheochromocytoma; Recurrent Renal Cell Cancer; Somatostatinoma; Stage III Neuroendocrine Carcinoma of the Skin; Stage IV Melanoma; Stage IV Non-small Cell Lung Cancer; Stage IV Renal Cell Cancer; Thyroid Gland Medullary Carcinoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Gastrinoma; Glucagonoma; Insulinoma; Pheochromocytoma; Carcinoma, Islet Cell; Melanoma; Carcinoma, Merkel Cell; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Somatostatinoma; Carcinoma, Medullary | interventions — Everolimus; vatalanib; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): See Detailed Description
  Interventions: Drug: everolimus; Drug: vatalanib; Other: pharmacological study; Other: laboratory biomarker analysis; Procedure: dynamic contrast-enhanced magnetic resonance imaging; Procedure: ultrasound imaging

INTERVENTIONS:
Drug: everolimus — Given orally
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Drug: vatalanib — Given orally
  Other Names: CGP-79787; PTK787/ZK 222584
Other: pharmacological study — Correlative study (Cohort IIA only)
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative study (Cohorts IIA and IIB)
Procedure: dynamic contrast-enhanced magnetic resonance imaging — Correlative study (Cohort IIA only)
  Other Names: DCE-MRI
Procedure: ultrasound imaging — Correlative study (Cohorts IIA and IIB)
  Other Names: ultrasonography; ultrasound; ultrasound test

SUMMARY:
RATIONALE: Everolimus and vatalanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving everolimus together with vatalanib may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of everolimus and vatalanib in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the dose limiting toxicity (DLT) and maximally tolerated dose (MTD) of RAD001 and once daily PTK787 when given in combination. (Cohort IA) II. To describe the toxicities associated with the combination of RAD001 and once daily PTK787. (Cohort IA) III. To evaluate the therapeutic antitumor activity of the combination of once daily PTK787 with RAD001. (Cohort IA) IV. To determine the dose limiting toxicity (DLT) and maximally tolerated dose (MTD) of RAD001 and twice daily PTK787 when given in combination. (Cohort IB) V. To describe the toxicities associated with the combination of RAD001 and twice daily PTK787. (Cohort IB) VI. To evaluate the therapeutic antitumor activity of the combination of twice daily PTK787 with RAD001. (Cohort IB) VII. To determine the MTD-Recommended Phase 2 Dose (RP2D) based on the MTD for Cohorts IA and IB. (Cohorts IA & IB) VIII. To investigate the biological activity of the combination of PTK787 with RAD001 at the MTD-RP2D. (Cohort II) IX. To evaluate the therapeutic antitumor activity of the combination of PTK787 with RAD001 at the MTD-RP2D. (Cohort II) X. To evaluate pharmacogenetic, metabolic and clinical markers that may predict for hypertension induced by anti-VEGF therapy. (Cohort II) XI. To obtain pilot data on efficacy outcomes in patients with metastatic kidney cancer, neuroendocrine cancer, NSCLC or melanoma. (Cohort II)

OUTLINE:

Patients are assigned to 1 of 4 cohorts, according to their disease (cohort IA, IB, or IIA [any histopathologic diagnosis] vs cohort IIB [metastatic kidney cancer, neuroendocrine cancer, melanoma, or non-small cell lung cancer). Patients are initially enrolled into cohorts IA and IB until the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) are determined. Once the MTD/RP2D of everolimus and vatalanib are determined, subsequent patients are enrolled and treated in expansion cohorts IIA or IIB.

Cohorts 1A or 1B (dose escalation cohorts; closed to enrollment as of 12/6/06): Patients receive oral vatalanib once (cohort 1A) or twice (cohort 1B) daily on days 1-28 and oral everolimus once daily on days 15-28 of course 1. For all subsequent courses, patients receive oral vatalanib once (cohort 1A) or twice (cohort 1B) daily and oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohort IIA (expansion cohort treated at the MTD/RP2D): Patients receive oral everolimus once daily for 14 days followed by a 7-day rest period. Patients then receive oral vatalanib twice daily on days 1-28 and oral everolimus once daily on days 15-28 of course 1. For all subsequent courses, patients receive oral vatalanib twice daily and oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohort IIB (expansion cohort treated at the MTD/RP2D): Patients receive oral vatalanib twice daily on days 1-28 and oral everolimus once daily on days 15-28 of course 1. For all subsequent courses, patients receive oral vatalanib twice daily and oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of cancer that is now unresectable (solid tumors, excluding lymphoma)
* Ability to provide informed consent
* Willingness to return to Mayo Clinic Rochester for follow up
* Life expectancy >= 12 weeks
* Prior anti-VEGF therapy allowed
* Cohort IIA: Patients meeting other eligibility criteria, regardless of histopathologic diagnosis; tumor that is amenable to biopsy; willingness to provide blood specimens, undergo DCE-MRI, and undergo brachial artery ultrasound measurements as required by the protocol
* The following laboratory values obtained =< 14 days prior to registration:

Negative for proteinuria based on dip stick reading OR, if documentation of +1 result for protein on dip stick reading, then total urinary protein =< 500 mg and measured creatinine clearance (CrCl) >= 50 mL/min from a 24-hour urine collection

* Cohort IIB: Patients meeting other eligibility criteria AND with pathologic diagnosis of metastatic kidney cancer, neuroendocrine carcinoma, melanoma, and NSCLC; willingness to provide blood specimens required and undergo brachial artery ultrasound measurements
* The following laboratory values obtained =< 14 days prior to registration:

ANC >= 1500/uL; Hgb >= 9 g/dL; PLT >= 100,000/uL; Total bilirubin =< 1.5 x upper limit of normal (ULN); AST =< 3 x ULN or AST =< 5 x ULN if liver involvement; Creatinine =< 1.5 x ULN; INR =< 1.4 (Cohort IIA only)

Exclusion Criteria:

* Any of the following prior therapies: Full field radiation therapy =<4 weeks prior to registration or limited field radiation therapy =< 2 weeks prior to registration; Radiation to >30% of bone marrow; Major surgery (i.e., laparotomy) =< 4 weeks prior to registration; Minor surgery =< 2 weeks prior to registration
* New York Heart Association classification III or IV
* Uncontrolled hypertension, labile hypertension or history of poor compliance with antihypertensive medication
* Active, bleeding diathesis or on any anticoagulant except patients receiving heparin for deep venous thrombosis prophylaxis (not treatment)
* CNS metastases or seizure disorder
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-FDA-approved indication and in the context of a research investigation
* Any concurrent severe and/or uncontrolled medical conditions which could compromise participation or pose as unnecessary risk to the patient in the study, including, but not limited, to the following: Unstable angina; Myocardial infarction =< 6 months prior to registration; Serious uncontrolled cardiac arrhythmia; Uncontrolled diabetes
* Any concurrent severe and/or uncontrolled medical conditions which could compromise participation or pose as unnecessary risk to the patient in the study, including, but not limited, to the following: Interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung; QTc > 500 msec; Patients who require chronic treatment with PPI or H2 antagonist
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK787/ZK 222584 (i.e., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the tablets)
* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Chemotherapy =< 3 weeks; Mitomycin C/nitrosoureas =< 6 weeks; Immunotherapy =< 2 weeks; Biologic therapy =< 2 weeks; Prior investigational therapy =< 4 weeks; Full field radiation therapy =< 4 weeks or limited field radiation therapy =< 2 weeks; Radiation to > 30% of bone marrow; Major surgery (i.e., laparotomy) =< 4 weeks; or Minor surgery =< 2 weeks prior to registration
* Any of the following: pregnant women; nursing women; men or women of childbearing potential who are unwilling to employ adequate barrier contraception
* Patients on whom DCE-MRI is contraindicated (e.g., presence of MRI-incompatible metallic implants or prosthetic heart valves, pacemakers, etc.) are ineligible
* ECOG performance status (PS) 3 or 4
* Treatment with medications listed in Appendix I for which no safer or more efficacious alternative is available
* Uncontrolled infection
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2004-12 (Actual); Primary Completion 2009-09-15 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of everolimus and vatalanib (Cohort I) (Closed to enrollment as of 12/6/06) | Up to 28 days post treatment cycle
Toxicity associated with everolimus and vatalanib (Cohort I) (Closed to enrollment as of 12/6/06) | Up to 28 days post treatment cycle
Therapeutic antitumor activity of everolimus and vatalanib (Cohort I) (Closed to enrollment as of 12/6/06) | Up to 28 days post treatment cycle
Recommended phase II dose (RP2D) of everolimus and vatalanib (Cohort I) (Closed to enrollment as of 12/6/06) | After MTD (maximum tolerate dose) is determined from Phase I
Biological activity and therapeutic antitumor activity of everolimus and vatalanib when given at the MTD/RPTD (Cohort II) | Post treatment cycle
Evaluation of pharmacogenetic, metabolic, and clinical markers that may predict hypertension induced by anti-VEGF therapy (Cohort II) | Day 1 and 14 of Cycle 1 of treatment
Efficacy outcomes in patients with metastatic kidney cancer, neuroendocrine carcinoma, non-small cell lung cancer, or melanoma (Cohort II) | Post treatment cycle with MTD outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Julian R. Molina, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States